CLINICAL TRIAL: NCT06377358
Title: Lipolysis of Visceral Reserve Fat Using Tecar Therapy: Anthropometric, Biochemical and NMR Imaging Study.
Brief Title: Study of Lipolysis of Visceral Reserve Fat Using Tecar Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAPENERGY MEDICAL, SL (Industry)
Collaborators: University of Malaga (Other); Alfonso X El Sabio University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEEAH CA31
Record Dates: First submitted 2024-02-27; First posted 2024-04-22 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Obesity, Visceral; Obesity; Endocrine
Keywords: Tecar Therapy; Fat; Inflammation; Adipokines
MeSH Terms: conditions — Obesity, Abdominal; Obesity; Platelet Glycoprotein IV Deficiency; Inflammation

STUDY DESIGN:
Intervention Model Description: Tecar Theraty was applied to 20 obese patients in order to assess the effect on the body fat loss, serum adipocytokines and imflammation. It was an interventional study in one group of patients. No controls. No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Obese patients (Experimental): Twenty obese patients treated by tecar therapy
  Interventions: Device: Tecar Therapy

INTERVENTIONS:
Device: Tecar Therapy — Tecar Therapy at 1Mhz radiofrequency by the use of a C-400 device. The duration of the treatment will be 5 weeks, where 10 sessions will be carried out, 2 per week

SUMMARY:
The Scope of this study is to assess the visceral and subcutaneous fat loss in patients having Tecar (Radiofrequency) Therapy and its effects on other anthropometric variables, adipokines and inflammation.

20 obese patients will be treated with Tecar Therapy (Radiofrequency). Each patient will have 4 active, automatic plates placed on the abdomen (200 cm2 per plate), two on the right side of the midline and two on the left side. Energy will be applied for 50 minutes, controlling the temperature. Subsequently, 15 minutes of Capacitive and Resistive manual electrodes will be applied to the abdomen, simultaneously, 20 minutes of Lymphatic Drainage placing one active plate in the foot and the other in the lumbo-dorsal area. Patients will be informed that they will only feel comfortable warmth. Five sessions will be applied from Monday to Friday resting Saturday and Sunday, for 2 weeks. Total 10 sessions.

Subcutaneous and visceral fat will be measured by MRI. Anthropometric variables (Body Mass Index, Waist to Hip ratio and skinfold) will be also measured.

Metabolic and inflammatory effects of the RF treatment will be evaluated measuring adipokines (Leptin, adiponectin and resistin) as well as citokines (IL-6, TNF-a and C reactive Protein).

Results will be analyzed using the SPSS statistics package. A Kolmogorov-Smirnov test will be applied, if the data behaves normally, parametric tests will be applied. If not, non-parametric tests will be performed. The differences between proportions will be analyzed using Fischer's exact test. The differences between the medians will be assessed using the Student's t-test for paired samples and independent samples.

DETAILED DESCRIPTION:
Radiofrequency (RF) is an inexpensive, virtually side-effect-free, well-tolerated method that reduces belly fat. RF is a form of high-frequency electromagnetic energy that works by heating tissues (Tecar Therapy). Its action in deeper tissues (subcutaneous layer) aims to increase cellular metabolism. When applied to tissues, RF generates oscillating magnetic fields that move electrically charged particles, producing heat in the tissues, and the amount of heat produced depends on the resistance (bioimpedance) of the target tissue. Electrical energy is converted into thermal energy. There is evidence of a transient RF effect on autonomic homeostasis with no known negative effects. This autonomic response to RF is reflected in a thermoregulatory vasomotor mechanism, in changes in chemoreceptor activity, and even in fluctuations in the renin-angiotensin system, responses related to the control of energy metabolism. The elevation of tissue temperature appears to be sufficient to activate the sympathetic branch of the Autonomic Nervous System, leading to the release of catecholamines (adrenaline and noradrenaline), which are the trigger to activate lipolysis. Lipolysis is the reversible biochemical process where triglyceride catabolism is stored. This process culminates in the generation of non-esterified fatty acids and glycerol. Fatty acids released into the bloodstream can be used as a substrate to produce energy.

Ex vivo human skin cultures after completion of the RF treatment series showed a significant effect on subcutaneous adipocytes. Adipocyte cells were observed to have altered morphology and increased expression of the apoptosis marker, APAF-1, suggesting that induced apoptosis is the mechanism of action. Adipocyte apoptosis results in the release of triglycerides from disintegrated cell membranes, but in a delayed and gradual manner, allowing for slow and safe elimination through the interstitial space, and subsequent lipid transport systems, lymphatic systems, and other metabolic functions. There was no evidence of necrosis or inflammatory changes observed in adipocytes after treatments with this new RF device.

Obesity causes an increase in adipose tissue and an increased infiltration of inflammatory cells into that tissue with a predominance of pro-inflammatory cytokines resulting in the development of a chronic low-intensity inflammatory state.

Adipocytolysis is a term used to describe the phenomena caused by non-surgical techniques (cytolytic methods) for the reduction of localized fat, in which lipids could be broken or solubilized through the partial or total rupture of adipocytes, destroying their plasma membrane.

Frequencies around 1 MHz are used, which are the ones that act most effectively on the cell, but with a high power, adjustable temperature and a treatment area greater than 200 cm2, which allows it to mechanically destroy the adipose cells, with greater effectiveness in the subcutaneous adipose tissue without damaging the skin. blood, vessels, nerves, or connective tissues. Lipids are gradually eliminated through the lymphatic system, reducing tissue volume.

This procedure has been used quite effectively in aesthetics to reduce subcutaneous fat.

Inflammation is an orderly sequence of events designed to maintain homeostasis of organs and tissues. Chronic inflammation that lasts a long time and is characterized by the presence of lymphocytes and macrophages and the proliferation of blood vessels and connective tissue. This is considered a characteristic feature of metabolic syndrome, characterized by the secretion of inflammatory adipokines usually from adipose tissue, such as leptin, interleukin (IL-6), tumor necrosis factor α (TNF-α), monocyte chemoattractant protein. 1 (MCP-1) and resistin. Obesity, which is a feature of metabolic syndrome, was associated with chronic inflammation in obese subjects. Several inflammatory indicators are linked to obesity and shed light on the associated health complications. Inflammatory indicators include IL-6 and C-reactive protein (CRP) as inflammatory markers and adiponectin as an anti-inflammatory marker.

Sustained inflammation is considered a major risk factor for developing many diseases, including cardiovascular disease, metabolic syndrome, diabetes, and cancer. As a risk factor, obesity predisposes to a pro-inflammatory state through the increase of inflammatory mediators IL-6 and TNF-α, and reduced levels of adiponectin, which has a totally anti-inflammatory function. The inflammatory state followed by vascular and endothelial dysfunction is characterized by a decrease in nitric oxide and an increase in reactive oxygen species leading to oxidative stress. Both states of oxidative stress and inflammation initiate atherosclerosis, hypertension, alteration of metabolic markers, and thus major adverse cardiovascular events. Hence the importance of studying these markers before and after treatment.

RF treatment induces an increase in the apoptotic index in adipocytes 1 hour after RF treatment. This is accompanied by a maximum temperature of 45°C in the grease layer. Skin surface temperatures remain substantially lower than fat temperatures.

While computed tomography (CT) is the most commonly used imaging modality for measuring abdominal fat, magnetic resonance imaging (MRI) has similar accuracy. An advantage of MRI is the absence of exposure to ionizing radiation, a limitation that restricts the use of CT in children and adolescents. In addition, the MRI method for quantifying abdominal adiposity is effective, allowing imaging within 5 minutes. Magnetic resonance imaging can provide reliable and good quality images for visceral and subcutaneous quantification.

OBJECTIVES MAIN OBJECTIVE. To evaluate the effect of high-power resistive capacitive radiofrequency on the decrease of visceral and subcutaneous fat and changes in the lipid profile and glucaemia, serum adipokine and inflammation markers.

SIDE OBJECTIVES. To evaluate and the decrease in abdominal circumferente measured by anthropometric tape measure, Body Mass Index, Waist-to-Hip Ratio and skinfold before and after RF treatment.

METHODOLOGY At the inclusion visit, the patient will be given the information sheet and, if they agree, they will be asked to sign the informed consent. Once included in the study, they will be randomly assigned to one of the two study groups in order of consecutive inclusion.

The project has been aprroved by the Ethics Committee of the Autonomous University of Barcelona UAB.

Sample size Calculation The aim of this study was to assess the difference between a decrease in the diameter of the abdominal circumference in a group of women, before and after radiofrequency treatment. The aim is to be able to declare a difference of 2 points or more as significant, taking the SD from published research that gives around 8.0 with a confidence level of 95%, a power of 80% and a correlation coefficient of 0.70 between the values of abdominal circumference before and after treatment. These are taken from the article published by Duarte et al. in 2015, and the following results are obtained according to EPIDATA: 15 pairs of data will then be taken: Before and after the application of RF.

TREATMENT Each patient will have 4 active, automatic plates placed on the abdomen (200 cm2 per plate), two on the right side of the midline and two on the left side. Energy will be applied for 50 minutes, controlling the temperature. Subsequently, 15 minutes of Capacitive and Resistive manual electrodes will be applied to the abdomen, simultaneously, 20 minutes of Lymphatic Drainage placing one active plate in the foot and the other in the lumbo-dorsal area. Patients will be informed that they will only feel comfortable warmth. Five sessions will be applied from Monday to Friday resting Saturday and Sunday, for 2 weeks. Total 10 sessions.

MEASUREMENTS (Technical details for primary and secondary outcomes)

* The adipose tissue volumes (cm3) of each compartment were calculated by adding the relevant voxel counts and multiplying by the voxel dimensions in cubic centimeters (cm3). The volume of adipose tissue for the entire abdomen was calculated by multiplying the volumes of adipose tissue from each slice by the sum of the thickness of the slice (5 mm) and the distance between slices. This analysis provides a direct measurement of adipose tissue volume. Adipose tissue in grams is calculated from the following formula:
* Fat mass (g) = Adipose tissue volume cm3 x 0.66 g/cm3
* Body Mass Index is calculated as follows: Body Weight (Kg) ÷ Height (m2)
* Waist-to-Hip Ratio: According to World Health Organization guidelines, the waist should be measured at the midpoint between the last palpable rib and the top of the iliac crest (upper edge of the pelvis). The hip should be measured at the point of maximum circumference. Both measures should be taken immediately after the air in the lungs is exhaled. The caliper takes the thickness of the abdominal wall at 5 cm in an oblique line towards the navel on the right and left side.
* Subcutaneous and visceral fat: will be measured using, in addition to the MRI method, an Inbody electrical impedance equipment, before ant after treatment.
* The skinfold thickness will be measured with a calliper.
* Biochemical parameters: fasting blood will be drawn from the patients, to obtain serum and EDTA-plasma, frozen until Assays. Interlukin-6, Tumor Necrosis Factor-alpha, leptin, adiponectin, resistin and ultrasensitive C-reactive protein will be determined By ELISA by inmmuneassays.

STATISTICAL ANALYSIS The statistical analysis of the results will be performed using the Software Package for Social Sciences (SPSS 24.0.).

A Kolmogorov-Smirnov test will be applied, if the data behaves normally, parametric tests will be applied. If not, non-parametric tests will be performed.

The differences between proportions will be analyzed using Fischer's exact test. The differences between the medians will be assessed using the Student's t-test for paired samples and independent samples.

ELIGIBILITY:
Inclusion criteria:

* Men and women.
* Age from 20 to 80 years.
* Waist circumference > 102 cm in men and > 88 cm in women.
* BMI > 25 Kg/mt2.
* Visceral fat quantification > 9 (on a scale of 20).

Exclusion Criteria:

* Refusal to sign the informed consent.
* Pregnancy.
* Patients with metal prostheses.
* Presence of active infection.
* Patients with oncological history with chemotherapy treatments or radiotherapy.
* Presence of diabetes.
* Presence of metabolic disease.
* Presence of arterial hypertension.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodríguez Lastra, PhD, MD, Principal Investigator — Alfonso X El Sabio University
Locations (1):
- Inneo Terapia Despi, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araki E, Oyadomari S, Mori M. Impact of endoplasmic reticulum stress pathway on pancreatic beta-cells and diabetes mellitus. Exp Biol Med (Maywood). 2003 Nov;228(10):1213-7. doi: 10.1177/153537020322801018. PMID 14610263
- [Background] Badawi A, Klip A, Haddad P, Cole DE, Bailo BG, El-Sohemy A, Karmali M. Type 2 diabetes mellitus and inflammation: Prospects for biomarkers of risk and nutritional intervention. Diabetes Metab Syndr Obes. 2010 May 26;3:173-86. doi: 10.2147/dmsott.s9089. PMID 21437087
- [Background] Belenky I, Margulis A, Elman M, Bar-Yosef U, Paun SD. Exploring channeling optimized radiofrequency energy: a review of radiofrequency history and applications in esthetic fields. Adv Ther. 2012 Mar;29(3):249-66. doi: 10.1007/s12325-012-0004-1. Epub 2012 Feb 29. PMID 22382873
- [Background] Bjorntorp P. "Portal" adipose tissue as a generator of risk factors for cardiovascular disease and diabetes. Arteriosclerosis. 1990 Jul-Aug;10(4):493-6. No abstract available. PMID 2196039
- [Background] Chang SL, Huang YL, Lee MC, Chang CH, Lin YF, Cheng CY, Hu S. Long-term follow-up for noninvasive body contouring treatment in Asians. Lasers Med Sci. 2016 Feb;31(2):283-7. doi: 10.1007/s10103-015-1852-0. Epub 2015 Dec 29. PMID 26714982
- [Background] Duarte FO, Sene-Fiorese M, de Aquino Junior AE, da Silveira Campos RM, Masquio DC, Tock L, Garcia de Oliveira Duarte AC, Damaso AR, Bagnato VS, Parizotto NA. Can low-level laser therapy (LLLT) associated with an aerobic plus resistance training change the cardiometabolic risk in obese women? A placebo-controlled clinical trial. J Photochem Photobiol B. 2015 Dec;153:103-10. doi: 10.1016/j.jphotobiol.2015.08.026. Epub 2015 Sep 2. PMID 26398817
- [Background] Ellulu MS, Patimah I, Khaza'ai H, Rahmat A, Abed Y. Obesity and inflammation: the linking mechanism and the complications. Arch Med Sci. 2017 Jun;13(4):851-863. doi: 10.5114/aoms.2016.58928. Epub 2016 Mar 31. PMID 28721154
- [Background] Alexiades-Armenakas M, Dover JS, Arndt KA. Unipolar radiofrequency treatment to improve the appearance of cellulite. J Cosmet Laser Ther. 2008 Sep;10(3):148-53. doi: 10.1080/14764170802279651. PMID 18788033
- [Background] Eloi JC, Epifanio M, de Goncalves MM, Pellicioli A, Vieira PF, Dias HB, Bruscato N, Soder RB, Santana JC, Mouzaki M, Baldisserotto M. Quantification of Abdominal Fat in Obese and Healthy Adolescents Using 3 Tesla Magnetic Resonance Imaging and Free Software for Image Analysis. PLoS One. 2017 Jan 27;12(1):e0167625. doi: 10.1371/journal.pone.0167625. eCollection 2017. PMID 28129354
- [Background] Fritz K, Salavastru C, Gyurova M. Clinical evaluation of simultaneously applied monopolar radiofrequency and targeted pressure energy as a new method for noninvasive treatment of cellulite in postpubertal women. J Cosmet Dermatol. 2018 Jun;17(3):361-364. doi: 10.1111/jocd.12525. Epub 2018 Mar 9. PMID 29524305
- [Background] Gabai VL, Meriin AB, Yaglom JA, Wei JY, Mosser DD, Sherman MY. Suppression of stress kinase JNK is involved in HSP72-mediated protection of myogenic cells from transient energy deprivation. HSP72 alleviates the stewss-induced inhibition of JNK dephosphorylation. J Biol Chem. 2000 Dec 1;275(48):38088-94. doi: 10.1074/jbc.M006632200. PMID 10978340
- [Background] Janssen I, Heymsfield SB, Allison DB, Kotler DP, Ross R. Body mass index and waist circumference independently contribute to the prediction of nonabdominal, abdominal subcutaneous, and visceral fat. Am J Clin Nutr. 2002 Apr;75(4):683-8. doi: 10.1093/ajcn/75.4.683. PMID 11916754
- [Background] Janssen I, Katzmarzyk PT, Ross R. Waist circumference and not body mass index explains obesity-related health risk. Am J Clin Nutr. 2004 Mar;79(3):379-84. doi: 10.1093/ajcn/79.3.379. PMID 14985210
- [Background] Kaplan H, Gat A. Clinical and histopathological results following TriPollar radiofrequency skin treatments. J Cosmet Laser Ther. 2009 Jun;11(2):78-84. doi: 10.1080/14764170902846227. PMID 19408182
- [Background] Klopfenstein BJ, Kim MS, Krisky CM, Szumowski J, Rooney WD, Purnell JQ. Comparison of 3 T MRI and CT for the measurement of visceral and subcutaneous adipose tissue in humans. Br J Radiol. 2012 Oct;85(1018):e826-30. doi: 10.1259/bjr/57987644. Epub 2012 Apr 18. PMID 22514099
- [Background] Kondo T, Sasaki K, Matsuyama R, Morino-Koga S, Adachi H, Suico MA, Kawashima J, Motoshima H, Furukawa N, Kai H, Araki E. Hyperthermia with mild electrical stimulation protects pancreatic beta-cells from cell stresses and apoptosis. Diabetes. 2012 Apr;61(4):838-47. doi: 10.2337/db11-1098. Epub 2012 Feb 23. PMID 22362176
- [Background] Maffeis C, Corciulo N, Livieri C, Rabbone I, Trifiro G, Falorni A, Guerraggio L, Peverelli P, Cuccarolo G, Bergamaschi G, Di Pietro M, Grezzani A. Waist circumference as a predictor of cardiovascular and metabolic risk factors in obese girls. Eur J Clin Nutr. 2003 Apr;57(4):566-72. doi: 10.1038/sj.ejcn.1601573. PMID 12700618
- [Background] Mazzoni D, Lin MJ, Dubin DP, Khorasani H. Review of non-invasive body contouring devices for fat reduction, skin tightening and muscle definition. Australas J Dermatol. 2019 Nov;60(4):278-283. doi: 10.1111/ajd.13090. Epub 2019 Jun 6. PMID 31168833
- [Background] Minami Y, Hohfeld J, Ohtsuka K, Hartl FU. Regulation of the heat-shock protein 70 reaction cycle by the mammalian DnaJ homolog, Hsp40. J Biol Chem. 1996 Aug 9;271(32):19617-24. doi: 10.1074/jbc.271.32.19617. PMID 8702658
- [Background] Moreno LA, Pineda I, Rodriguez G, Fleta J, Sarria A, Bueno M. Waist circumference for the screening of the metabolic syndrome in children. Acta Paediatr. 2002;91(12):1307-12. doi: 10.1080/08035250216112. PMID 12578286
- [Background] Morino S, Suico MA, Kondo T, Sekimoto E, Yano S, Matsuda T, Matsuno T, Shuto T, Araki E, Kai H. Mild electrical stimulation increases ubiquitinated proteins and Hsp72 in A549 cells via attenuation of proteasomal degradation. J Pharmacol Sci. 2008 Oct;108(2):222-6. doi: 10.1254/jphs.08180sc. Epub 2008 Oct 10. PMID 18845908
- [Background] Mulholland RS, Paul MD, Chalfoun C. Noninvasive body contouring with radiofrequency, ultrasound, cryolipolysis, and low-level laser therapy. Clin Plast Surg. 2011 Jul;38(3):503-20, vii-iii. doi: 10.1016/j.cps.2011.05.002. PMID 21824546
- [Background] Ohlson LO, Larsson B, Svardsudd K, Welin L, Eriksson H, Wilhelmsen L, Bjorntorp P, Tibblin G. The influence of body fat distribution on the incidence of diabetes mellitus. 13.5 years of follow-up of the participants in the study of men born in 1913. Diabetes. 1985 Oct;34(10):1055-8. doi: 10.2337/diab.34.10.1055. PMID 4043554
- [Background] Park HS, Lee JS, Huh SH, Seo JS, Choi EJ. Hsp72 functions as a natural inhibitory protein of c-Jun N-terminal kinase. EMBO J. 2001 Feb 1;20(3):446-56. doi: 10.1093/emboj/20.3.446. PMID 11157751
- [Background] Pereira JX, Cavalcante Y, Wanzeler de Oliveira R. The role of inflammation in adipocytolytic nonsurgical esthetic procedures for body contouring. Clin Cosmet Investig Dermatol. 2017 Feb 23;10:57-66. doi: 10.2147/CCID.S125580. eCollection 2017. PMID 28260937
- [Background] Pinto H. Local fat treatments: classification proposal. Adipocyte. 2015 Jun 26;5(1):22-6. doi: 10.1080/21623945.2015.1066534. eCollection 2016 Jan-Mar. PMID 27144093
- [Background] Pumprla J, Howorka K, Kolackova Z, Sovova E. Non-contact radiofrequency-induced reduction of subcutaneous abdominal fat correlates with initial cardiovascular autonomic balance and fat tissue hormones: safety analysis. F1000Res. 2015 Feb 20;4:49. doi: 10.12688/f1000research.5708.1. eCollection 2015. PMID 26069728
- [Background] Rexrode KM, Carey VJ, Hennekens CH, Walters EE, Colditz GA, Stampfer MJ, Willett WC, Manson JE. Abdominal adiposity and coronary heart disease in women. JAMA. 1998 Dec 2;280(21):1843-8. doi: 10.1001/jama.280.21.1843. PMID 9846779
- [Background] Ryden M, Arner P. Subcutaneous Adipocyte Lipolysis Contributes to Circulating Lipid Levels. Arterioscler Thromb Vasc Biol. 2017 Sep;37(9):1782-1787. doi: 10.1161/ATVBAHA.117.309759. Epub 2017 Jun 29. PMID 28663255
- [Background] Sharp FR, Massa SM, Swanson RA. Heat-shock protein protection. Trends Neurosci. 1999 Mar;22(3):97-9. doi: 10.1016/s0166-2236(98)01392-7. No abstract available. PMID 10199631
- [Background] Shinohara T, Takahashi N, Ooie T, Hara M, Shigematsu S, Nakagawa M, Yonemochi H, Saikawa T, Yoshimatsu H. Phosphatidylinositol 3-kinase-dependent activation of akt, an essential signal for hyperthermia-induced heat-shock protein 72, is attenuated in streptozotocin-induced diabetic heart. Diabetes. 2006 May;55(5):1307-15. doi: 10.2337/db05-0266. PMID 16644687
- [Background] Sugawara J, Kou S, Kokubo K, Kuroda A, Hashizume Y, Kobayashi S, Maegawa J, Satake T. Application for lower facial fat reduction and tightening by static type monopolar 1-MHz radio frequency for body contouring. Lasers Surg Med. 2017 Oct;49(8):750-755. doi: 10.1002/lsm.22676. Epub 2017 Apr 22. PMID 28432775
- [Background] van der Lugt C, Romero C, Ancona D, Al-Zarouni M, Perera J, Trelles MA. A multicenter study of cellulite treatment with a variable emission radio frequency system. Dermatol Ther. 2009 Jan-Feb;22(1):74-84. doi: 10.1111/j.1529-8019.2008.01218.x. PMID 19222519
- [Background] World Health Organization. Waist circumference and waist-hip ratio - Report of a WHO expert consultation, Geneva, 8-11 December 2008
- [Background] Wu B, Hunt C, Morimoto R. Structure and expression of the human gene encoding major heat shock protein HSP70. Mol Cell Biol. 1985 Feb;5(2):330-41. doi: 10.1128/mcb.5.2.330-341.1985. PMID 2858050
- [Derived] Rodriguez Lastra J, Kouser S. Reduction of Subcutaneous and Visceral Fat With the Use of Energy-Based Equipment With a High-Power Amplifying Effect Plus an Exercise Regimen. J Cosmet Dermatol. 2025 Oct;24(10):e70490. doi: 10.1111/jocd.70490. PMID 41059542

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obese Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Total 20 men (10) and women (10) aged 20 to 80 years, with waist circumference > 102 cm in men and > 88 cm in women, a BMI > 25 Kg/m2 and visceral fat quantification > 9 (on a scale of 20) have been recruited
Arm/Group | Obese Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 20
Visceral adipose Tissue (VAT) in grams (g) [Mean (Standard Deviation); unit: grams] | 3988 (1850)
Subcutaneous Fat Tissue (SFT) in g [Mean (Standard Deviation); unit: grams] | 9124 (2804)

OUTCOME MEASURES:

1. Primary Outcome: Visceral Fat Loss (cm3)
Description: Measurement of Visceral fat loss (cm3) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: cm3
Groups:
- 20 Obese Patients: Twenty obese patients treated by TECAR therapy
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
cm3 | -628 (103)

2. Primary Outcome: Visceral Fat Loss (g)
Description: Measurement of Visceral fat loss (g) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
grams | -565 (93)

3. Primary Outcome: Subcutaneous Fat Loss (cm3)
Description: Measurement of subcutaneous fat loss (cm3) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by tecar therapy Tecar Therapy
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
cm3 | -803 (492)

4. Primary Outcome: Subcutaneous Fat Loss (g)
Description: Measurement of subcutaneous fat loss (g) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients were treated by TECAR therapy.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
grams | -845 (433)

5. Primary Outcome: Tumor Necrosis Factor Alfa
Description: Changes in serum/plasma levels of Tumor Necrosis Factor alfa (pg/mL) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients were treated by TECAR therapy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
pg/mL | 0.70 (2.5)

6. Primary Outcome: Interleukin 6 Levels
Description: Changes in serum/plasma levels of Interleukin 6 (pg/mL) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
pg/mL | -0.53 (2.2)

7. Primary Outcome: C Reactive Protein Levels
Description: Changes in serum/plasma C reactive Protein (mg/L) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
mg/L | 0.12 (3.14)

8. Primary Outcome: Leptin Levels
Description: Changes in serum/plasma levels of leptin after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
ng/mL | -7.33 (7.28)

9. Primary Outcome: Adiponectin Levels
Description: Changes in serum/plasma levels of adiponectin after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
ng/mL | -296.9 (1023.8)

10. Primary Outcome: Resistin Levels
Description: Changes in serum/plasma levels of resistin after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
ng/mL | -0.19 (1.21)

11. Primary Outcome: Total Cholesterol Changes
Description: Measurement of serum total cholesterol (mg/dL) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
mg/dL | -11.8 (16.8)

12. Primary Outcome: Total Triglycerides Changes
Description: Measurement of serum total triglycerides (mg/dL) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
mg/dL | -15.6 (46)

13. Primary Outcome: LDL Cholesterol Changes
Description: Measurement of serum LDL Cholesterol (mg/dL) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
mg/dL | -6.15 (21.6)

14. Primary Outcome: HDL Cholesterol Changes
Description: Measurement of serum HDL Cholesterol (mg/dL) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
mg/dL | -2.6 (5.47)

15. Primary Outcome: Glucose
Description: Measurement of Glucose (mg/dL) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
mg/dL | -3.5 (6.83)

16. Secondary Outcome: Body Mass Index Loss
Description: Measurement of Body Mass Index loss (Kg/m2) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
kg/m2 | 0 (2)

17. Secondary Outcome: Waist to Hip Ratio (WHR-unitless) Loss
Description: Measurement of the WHR loss after the Tecar Therapy treatment. It is calculated by dividing waist circumference by hip circumference. It is a unitless measure indicating fat distribution, with lower values reflecting reduced abdominal fat.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
unitless | -0.02 (0.05)

18. Secondary Outcome: Skinfold Thickness (mm)
Description: Measurement of the Skinfold Thickness (mm) after Tecar Therapy treatment.
Time Frame: 3 months
Population: Twenty obese patients treated by TECAR therapy
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 20 Obese Patients
Number analyzed (Participants) | 20
mm | -1.85 (2.36)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: No Serious Adverse Events or All-Cause Mortality occurred during the study
Arm/Group | Obese Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese Patients (N=20)
Erythema (Skin and subcutaneous tissue disorders) | 4 (10) — Redness

LIMITATIONS AND CAVEATS:
The limited sample size of this study, with only 20 participants recruited, represents a key limitation. Additionally, financial constraints posed a challenge, as covering the costs of MRI scans and blood analyses for a larger sample was not feasible

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT06377358/Prot_SAP_002.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT06377358/ICF_001.pdf